CLINICAL TRIAL: NCT02512081
Title: "The Lived Experience of Investigations in Sciatica"
Brief Title: "The Lived Experience of Investigations for Sciatica"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Collaborators: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: UOS-2307-CR
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-07

CONDITIONS: Sciatica
Keywords: Sciatica; Patient Experience; Investigations; Qualitative Research
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention applied — No intervention applied

SUMMARY:
This will be an exploratory study, using semi-structured interviews to explore patients' experiences of undergoing investigations for Sciatica (leg pain referred from the lower back). Interviews will be analysed based on an Interpretative Phenomenological Approach (IPA).The end product of analysis will be a detailed account of patients' experiences supported by direct quotes.The intention is that this account will help health-care providers to understand patients' experiences and to plan and provide Sciatica care that is effective, evidence based and acceptable to patients.

DETAILED DESCRIPTION:
Sciatica (leg pain referred from the lower back) is a common problem that causes significant pain and disability. Many patients experience lasting symptoms that do not respond to pain relief or physiotherapy. This group of patients are commonly managed by Spinal Specialists who help determine the best treatment approach and consider if investigations are required. In the United Kingdom (UK), clinical guidelines suggest that imaging for Sciatica is only appropriate for patients who are considered likely to need surgery or when the cause is suspected to be serious such as cancer or infection. Patients who do not meet the criteria for investigations express frustration when clinical tests and opinion alone are used to diagnose and treat Sciatica. Some patients are unable to accept that investigations are not required and loose confidence in treatment. If Sciatica is to be managed effectively, the treatment offered must be acceptable to and successfully negotiated with patients.

Little research is currently available regarding patients' expectations or experiences of undergoing investigations for Sciatica. The aim of this study is to explore the experience of patients who have undergone investigations for Sciatica, to gain an understanding of how patients experience investigations as part of their overall management of Sciatica.This study specifically explores the experiences of patients whose Sciatica is likely to be caused by nerve root involvement.

This study will be exploratory, based on an Interpretative Phenomenological Approach (IPA). Up to 15 patients who have undergone investigations for Sciatica will be interviewed using a semi-structured format. Patients will be recruited from one National Health Service (NHS) Trust on the South Coast of England. Interviews will be audio-recorded, transcribed verbatim and analysed thematically, based on an IPA approach. The end product of analysis will be a detailed account of patient's experience of investigations, supported by direct quotes. The intention is that this account will help health-care providers to understand patients' experiences and to plan and provide Sciatica care that is effective, evidence based and acceptable to patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Sciatica (of likely nerve root origin) Have undergone investigations for Sciatica and received results in past 6 weeks Patients who are able to read, write and understand English language instructions

Exclusion Criteria:

Previous spinal surgery Sciatica caused by sinister pathology or Cauda Equina Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged over 18 years) with a clinical diagnosis of 'Sciatica of likely nerve root origin' who have undergone investigations as part of their conservative management and received results in the past 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Patient Experience | Within 6 weeks of receiving investigation results for sciatica
  Patient experience gained through semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Roberts, Associate Professor, Study Chair — University of Southampton